CLINICAL TRIAL: NCT03676803
Title: Effect of Spice Consumption on the Microbiome in Healthy Subjects: A Pilot Study
Brief Title: Effect of Spice Consumption on the Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor and Chief, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB#17-000617
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Microbiota
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed spices intervention group (Experimental): healthy participants consume a capsule containing 5 g of mixed spices at culinary dose
  Interventions: Other: mixed spices
- placebo group (Placebo Comparator): healthy participants consume placebo capsule containing 5 g of maltodextrin
  Interventions: Other: placebo capsule containing 5 g of maltodextrin

INTERVENTIONS:
Other: mixed spices — All spices in the spice mixture capsules contains 1g or 20% cinnamon, 1.5g or 30% oregano, 1.5g or 30% ginger, 0.85g or 17% black pepper, 0.15g or or 3% cayenne pepper for a total of 5.0g spice mixture. They are identical to herbs and spices sold in grocery stores for human consumption.
  Arms: Mixed spices intervention group
Other: placebo capsule containing 5 g of maltodextrin — placebo capsule containing 5 g of maltodextrin
  Arms: placebo group

SUMMARY:
Several human intervention studies have also been performed that demonstrated beneficial effects of high polyphenol fruits and vegetable on the intestinal microbiome. No information is available about the effect of spice consumption on the gut microbiome.

This proposed pilot study will assess the ability of daily consumption of 5 grams of mixed spices to alter the gut microbiome composition compared to placebo in a free-living population.

DETAILED DESCRIPTION:
This will be a randomized, double-blinded, placebo controlled design. Thirty-one subjects will be randomized to consume either 5 grams of mixed spice or matched placebo for 2 weeks in random sequence. At baseline and week 2, fasting blood, urine and stool will be collected. In addition body weight and composition will be determined and questionnaires and 3-day food record will be completed. Stool samples will be collected for sequencing of bacterial DNA to determine changes in the microbiota. The objective of the proposed pilot study is to determine whether intake of spice per day will alter the intestinal microflora leading to an increase in formation of short chain fatty acids.

Subjects will be assigned an enrollment number after signing the informed consent form approved by the UCLA Medical Internal Review Board. Eligible subjects will be enrolled into the study upon completion of screening evaluations, which include a physical exam, complete medical history, and blood drawing.

This study will be conducted in healthy free-living subjects (18-65 years). Subjects consume 5 gram mixed spices or placebo capsules daily for 2 weeks. Subjects will be instructed to eat a beige diet (low fiber<10g and low polyphenols <3 servings of polyphenol rich fruit/vegetables per day) during the entire study period. Participants will meet with the dietitian for instructions on eating a beige diet and will be instructed to follow the diet during the entirety of the study.

All spices in the spice mixture capsules contains 1g or 20% cinnamon, 1.5g or 30% oregano, 1.5g or 30% ginger, 0.85g or 17% black pepper, 0.15g or or 3% cayenne pepper for a total of 5.0g spice mixture - identical to herbs and spices sold in grocery stores for human consumption. There are no known safety issues with any of the ingredients.

Placebo capsules will contain maltodextrin equivalent to mixed spice blend.

Body weight will be measured on an uncarpeted surface on a scale (Detecto-Medic; Detecto-Scales; Brooklyn, NY) while wearing no shoes and after an overnight fast. Height is measured without shoes with a stadiometer (Detecto-Medic; Detecto-Scales; Brooklyn, NY) and recorded to the nearest 0.1 cm. Body composition will be measured using the Tanita-BC418 body-fat analyzer (Tanita Corp., Tokyo, Japan).

ELIGIBILITY:
Inclusion Criteria:

* Healthy human adults age 18-65 years old
* Typically consume low fiber/polyphenol diet (beige diet)-

Exclusion Criteria:

* Eating a high fiber/polyphenol diet or taking any medication or dietary supplement which interfere with the absorption of polyphenols.
* History of gastrointestinal surgery, diabetes mellitus, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP >160mmHg, diastolic BP > 95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
* Pregnant or breastfeeding
* Currently uses tobacco products.
* Is unable or unwilling to comply with the study protocol.
* Frequently using prebiotics, probiotics, yogurt, and/or any fiber supplements
* Allergy or sensitivity to spices. Subjects will be excluded if there is a prior history of such sensitivity. Since these foods are commonly eaten and allergies are rare, subjects should be aware of this sensitivity prior to entering the study. To determine this, a positive history of spices ingestion without incident will be requested. In addition, any subject with a history of allergy or anaphylaxis of any kind will be excluded
* Taking antibiotics or laxatives within the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — Center for Human Nutrition, UCLA David Geffen School of Medicine
Locations (1):
- UCLA Center for Human Nutrition, 900 Veteran Ave., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Interested participants who responded to the approved flyers called the research site and a coordinate conducted a screening by utilizing a screening script. Initial eligibility was determined by a telephone conversation. Eligible subjects were scheduled for a screen visit.
Pre-assignment Details: After one week run-in period, thirty-one participants were enrolled and randomized into mixed-spices intervention group and placebo group. All have completed the two-week intervention study.
Groups:
- Mixed Spices Intervention Group: Healthy participants consume a capsule containing 5 g of mixed spices at culinary dose
  Mixed spice capsules contain 1 g cinnamon, 1.5 g oregano, 1.5 g ginger, 0.85g black pepper and 0.15g cayenne pepper for a total of 5.0 g. They are identical to herbs and spices sold in grocery stores for human consumption.
- Placebo Group: Healthy participants consume placebo capsule containing 5 g of maltodextrin
  Placebo capsules contain 5 g maltodextrin.
Period: Overall Study
Arm/Group | Mixed Spices Intervention Group | Placebo Group
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mixed Spices Intervention Group: Healthy participants consume a capsule containing 5 g of mixed spices at culinary dose
  Mixed spice capsules contain 1 g cinnamon, 1.5 g oregano, 1.5 g ginger, 0.85g black pepper and 0.15g cayenne pepper for a total of 5.0 g.
- Total: Total of all reporting groups
Arm/Group | Mixed Spices Intervention Group | Placebo Group | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (12.2) | 35.6 (13.7) | 35.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3 | 1 | 4
  White | 7 | 9 | 16
  Asian | 3 | 3 | 6
  Multi-racial | 1 | 3 | 4
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (6.8) | 26.7 (4.4) | 27.5 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Microbial Phylum Abundance (% of Total) Between Spice and Placebo
Description: Change in microbial phylum abundance (% of total) between spice and placebo after two week intervention
Time Frame: 2-weeks
Population: Data from one participant from spice group and one from placebo group were excluded due to non-compliance with the protocol.
Measure: Mean (Standard Deviation); unit: percentage of total bacteria
Groups:
- Mixed Spices Intervention Group: Healthy participants consume a capsule containing 5 g of mixed spices daily for 2 weeks
- Placebo Group: Healthy participants consumed placebo capsules daily for 2 weeks.
Arm/Group | Mixed Spices Intervention Group | Placebo Group
Number analyzed (Participants) | 14 | 15
percentage of total bacteria
  Phylum Firmicutes at Baseline | 65.1 (10.5) | 65.9 (9.2)
  Phylum Firmicutes at Week 2 | 58.7 (13.3) | 70.1 (8.9)
  Phylum Bacteroidetes at Baseline | 28.2 (11.9) | 25.9 (7.9)
  Phylum Bacteroidetes at Week 2 | 33.6 (13.5) | 22.6 (8.4)
Statistical Analysis 1: Comparison: Mixed Spices Intervention Group vs Placebo Group; Comparison was made to 2 weeks minus baseline changes in phylum Firmicutes abundance between groups; Test type: Other; p = 0.033, ANOVA — p<0.05 was defined as significant; Mean Difference (Final Values) = 10.6
Statistical Analysis 2: Comparison: Mixed Spices Intervention Group vs Placebo Group; Comparison was made to 2 weeks minus baseline changes in phylum Bacteroidetes abundance between groups; Test type: Other; p = 0.097, ANOVA — p<0.05 was defined as significant; Mean Difference (Final Values) = 8.7

2. Secondary Outcome: Change From Baseline in Short-chain Fatty Acids (SCFAs) at 2 Weeks
Description: Change from baseline in total SCFAs including acetate, propionate, butyrate and valerate in response to mixed-spice intervention for 2 weeks. SCFAs were measured in dry fecal sample determined as micromole per gram of dry weight.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: micromole/g
Groups:
- Mixed Spices Intervention Group: Healthy participants consumed 5 g of mixed spices daily for 2 weeks
- Placebo Group: Healthy participants consumed placebo capsules containing 5 g of maltodextrin daily for 2 weeks
Arm/Group | Mixed Spices Intervention Group | Placebo Group
Number analyzed (Participants) | 14 | 15
micromole/g
  Total SCFAs at Baseline | 595.6 (311.6) | 678.0 (328.1)
  Total SCFAs at week 2 | 681.6 (333.2) | 733.7 (443.8)
Statistical Analysis 1: Comparison: Mixed Spices Intervention Group; Comparison was made to 2 weeks minus baseline in mixed spices intervention group; Test type: Other; p = 0.49, t-test, 2 sided; Mean Difference (Final Values) = 86.0
Statistical Analysis 2: Comparison: Placebo Group; Comparison was made to 2 weeks minus baseline in placebo group; Test type: Other; p = 0.53, t-test, 2 sided; Mean Difference (Final Values) = 55.7

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Mixed Spices Intervention Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 2/15 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mixed Spices Intervention Group (N=15) | Placebo Group (N=16)
stomach discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) — Bloating, nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT03676803/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT03676803/SAP_001.pdf